CLINICAL TRIAL: NCT00834093
Title: A Phase II Study of Epstein-Barr Virus-Specific Immunotherapy for Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Glenn J. Hanna, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-292; R21CA132279-01A1 (NIH)
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Epstein-Barr Virus; NPC; EBV; immunotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Epstein-Barr Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EBV-stimulated cytotoxic T-lymphocyte (EBV-CTL) Immunotherapy (Experimental): Eligible participants underwent a blood draw to obtain peripheral blood mononuclear cells (PBMCs) used for preparation of the immunotherapy product [estimated preparation time 14-16 weeks]. Participants received palliative chemotherapy for NPC as standard of care during the period required for T-cell production. Participants who achieved a partial response or better while receiving palliative chemotherapy continued to receive chemotherapy for 3 to 6 cycles and were only eligible for immunotherapy when progressive disease (PD) was confirmed. Each participant received a minimum of 2 EBV-CTL infusions, given 2 weeks apart, at doses of 1x108 cells/m2. A 3rd infusion was offered to participants 8-12 weeks after the 2nd infusion based on response, tolerability and sufficient immunotherapy product reserves.
  Interventions: Biological: Epstein-Barr Virus Specific Immunotherapy

INTERVENTIONS:
Biological: Epstein-Barr Virus Specific Immunotherapy
  Other Names: Cell based vaccine

SUMMARY:
The purpose of this research study is to determine how effective and how safe it is to give an Epstein-Barr Virus (EBV) immunotherapy product to participants with nasopharyngeal carcinoma (NPC) associated with EBV that has come back or spread to other parts of the participant's body. This is phase II study with the aim of establishing a baseline of efficacy.

DETAILED DESCRIPTION:
The study follows a pilot study optimizing and refining the manufacturing process, streamlining logistics (eg infusion protocol, enrolling out-of-town patients), increasing the cell dose, defining optimal patient eligibility, and improving monitoring for patients. Eligible participants will undergo a blood draw to obtain peripheral blood mononuclear cells (PBMCs) used for preparation of the immunotherapy product [estimated time 14-16 weeks]. Participants' PBMCs will be isolated by density centrifugation from peripheral blood and then infected with EBV to generate EBV-transformed B-lymphoblastoid cell lines (LCLs). LCLs will be irradiated and then used to stimulate autologous T cells, yielding an EBV-specific, autologous T cell product.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven NPC of an WHO grade, associated with EBV infection documented by the presence of EBER expression by in situ hybridization in the tumor. Positive EBER staining from another institution must be confirmed by pathology review at Brigham and Women's Hospital. Other confirmation of EBV-associated disease is acceptable, such as EBV DNA in situ hybridization, if EBER analysis is not adequate
* Incurable NPC
* Recovery from toxicity from any prior NPC therapy to grade 1 or better
* 18 years of age or older
* Evaluable or measurable disease, according to modified RECIST
* ECOG Performance Status of 0 or 1
* Adequate bone marrow, liver and renal function as outlined in protocol

Exclusion Criteria:

* Radiotherapy for primary NPC within 8 weeks of enrollment, or radiotherapy for any other reason within 6 weeks
* Chemotherapy for NPC within 2 weeks of enrollment
* Other cancer in the past 5 years, except for carcinoma in situ of the cervix or bladder, or non-melanomatous skin cancer
* Uncontrolled central nervous system metastases
* Active hepatitis, known HIV, or other condition that requires immunosuppressive therapy, including current use of high dose systemic corticosteroids
* Autoimmune disease, such as systemic lupus erythematosis or rheumatoid arthritis, that is active and requires current immunosuppressive therapy
* Active uncontrolled serious infection
* Women of child-bearing potential who have a positive pregnancy test or are breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2012-03 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Hanna, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No
There are no plans to share IPD. Cumulative results will be posted and published.

REFERENCES:
- [Result] Huang J, Fogg M, Wirth LJ, Daley H, Ritz J, Posner MR, Wang FC, Lorch JH. Epstein-Barr virus-specific adoptive immunotherapy for recurrent, metastatic nasopharyngeal carcinoma. Cancer. 2017 Jul 15;123(14):2642-2650. doi: 10.1002/cncr.30541. Epub 2017 Feb 21. PMID 28222215

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled from April 2009 to July 2011.
Period: Overall Study
Arm/Group | EBV-stimulated Cytotoxic T-lymphocyte (EBV-CTL) Immunotherapy
Started | 18
Eligible and Treated | 13
Completed | 10
Not Completed | 8
Not completed — Progressive Disease | 3
Not completed — Withdrawal by subject or MD Decision | 5

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of eligible and treated participants.
Arm/Group | EBV-stimulated Cytotoxic T-lymphocyte (EBV-CTL) Immunotherapy
Number analyzed (Participants) | 18
Age, Continuous [Mean (Full Range); unit: years] | 49 [20 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria on treatment. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Restaging scans were performed every 8 weeks on treatment up to 20 weeks.
Population: The analysis dataset is comprised of eligible and treated participants.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- EBV-stimulated Cytotoxic T-lymphocyte (EBV-CTL) Immunotherapy: Eligible participants undergo a blood draw to obtain peripheral blood mononuclear cells (PBMCs) used for preparation of the immunotherapy product [estimated time 14-16 weeks]. Participants receive palliative chemotherapy for NPC as standard of care during the period required for T-cell production. Each participant receives a minimum of 2 T-cell product infusions, given 2 weeks apart. A 3rd infusion may be given 8-12 weeks later based on response, tolerability and sufficient immunotherapy product reserves.Eligible participants underwent a blood draw to obtain peripheral blood mononuclear cells (PBMCs) used for preparation of the immunotherapy product [estimated preparation time 14-16 weeks]. Participants received palliative chemotherapy for NPC as standard of care during the period required for T-cell production. Participants who achieved a partial response or better while receiving palliative chemotherapy continued to receive chemotherapy for 3 to 6 cycles and were only eligible for immunotherapy when progressive disease (PD) was confirmed. Each participant received a minimum of 2 EBV-CTL infusions, given 2 weeks apart, at doses of 1x108 cells/m2. A 3rd infusion was offered to participants 8-12 weeks after the 2nd infusion based on response, tolerability and sufficient immunotherapy product reserves.
Arm/Group | EBV-stimulated Cytotoxic T-lymphocyte (EBV-CTL) Immunotherapy
Number analyzed (Participants) | 13
percentage of participants | 0.0 [0.0 to 20.6]

2. Secondary Outcome: Time to Progression (TTP)
Description: TTP estimated using the Kaplan-Meier method is defined as the duration of time from registration to documented first observation of progressive disease (PD), or censored at date last known progression-free. Based on RECIST 1.1, radiographic PD is defined as at least a 20% increase in the sum of the longest diameter (LD) for all target lesions (up to 10), taking as reference the smallest sum LD since beginning treatment or the appearance of one or more new lesions. For non-target lesions, PD is the appearance of one or more new lesions and/or unequivocal progression of existing lesions.
Time Frame: Restaging scans were performed every 8 weeks until PD. Follow-up duration was up to 92 months.
Population: The analysis dataset is comprised of eligible and treated participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | EBV-stimulated Cytotoxic T-lymphocyte (EBV-CTL) Immunotherapy
Number analyzed (Participants) | 13
months | 7.9 [6.7 to 9.9]

3. Secondary Outcome: Number of Participants With Grade 1-2 Fatigue Adverse Events," as Accurate and Appropriate
Description: All grade 1-2 fatigue adverse events (AE) with any treatment attribution as reported on case report forms were counted. The number of participants experiencing at least one grade 1-2 fatigue AE during the time of observation.
Time Frame: Adverse events were assessed after each infusion treatment. Treatment duration was up to 66 months.
Population: The analysis dataset is comprised of eligible and treated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | EBV-stimulated Cytotoxic T-lymphocyte (EBV-CTL) Immunotherapy
Number analyzed (Participants) | 13
Participants | 9

4. Secondary Outcome: Overall Survival (OS)
Description: OS estimated using the Kaplan-Meier (KM) method is defined as the time from registration to death, or censored at the date last known alive.
Time Frame: Participants were followed for survival per institutional practice until death or lost-to-follow-up. Follow-up duration was up to 92 months.
Population: The analysis dataset is comprised of eligible and treated participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | EBV-stimulated Cytotoxic T-lymphocyte (EBV-CTL) Immunotherapy
Number analyzed (Participants) | 13
months | 25.0 [6.0 to 28.2]

ADVERSE EVENTS:
Time Frame: Serious Adverse Events and Other Adverse Events were assessed throughout the treatment duration for up to 66 months. All-Cause Mortality was monitored until death or when lost-to-follow-up, for up to 92 months.
Description: Serious AEs were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv3. All remaining events regardless of treatment attribution were classified as Other AEs. Maximum grade toxicity by type for a patient over time was calculated. No further data is available to specify classification of other beyond the general term.
Arm/Group | EBV-stimulated Cytotoxic T-lymphocyte (EBV-CTL) Immunotherapy
All-Cause Mortality (participants affected / at risk) | 8/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 13/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EBV-stimulated Cytotoxic T-lymphocyte (EBV-CTL) Immunotherapy (N=13)
Infection w/ unk ANC conjunctiva (Infections and infestations) | 1
Otitis, external ear (non-infectious) (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Ocular-other (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Dry mouth (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Abdomen, pain (Gastrointestinal disorders) | 1
Dental/teeth/peridontal, pain (Gastrointestinal disorders) | 1
Stomach, pain (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 9
Constitutional, other (General disorders) | 1
Pain-other (General disorders) | 5
Flu-like syndrome (General disorders) | 2
Infection Gr0-2 neut, sinus (Infections and infestations) | 1
Infection-other (Infections and infestations) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Nonneuropathic lower extr muscle weak (Musculoskeletal and connective tissue disorders) | 1
Back, pain (Musculoskeletal and connective tissue disorders) | 6
Bone, pain (Musculoskeletal and connective tissue disorders) | 1
Joint, pain (Musculoskeletal and connective tissue disorders) | 1
Taste disturbance (Nervous system disorders) | 2
Neuropathy-sensory (Nervous system disorders) | 5
Neurologic-other (Nervous system disorders) | 1
Head/headache (Nervous system disorders) | 2
Urinary frequency/urgency (Renal and urinary disorders) | 1
Respiratory tract hemorrhage NOS (Respiratory, thoracic and mediastinal disorders) | 1
Throat/pharynx/larynx, pain (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 1
Nail changes (Skin and subcutaneous tissue disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 3
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1
Skin-other (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
The number of evaluable participants did not meet protocol objectives (n=13 versus target n=18).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No